





# Formulaire d'information à l'étude DE FACTO 2 « Etude interventionnelle sur les DEterminants et Facteurs de l'ACtivité physique après les Traitements en Oncologie »

Promoteur de l'étude : Université Sorbonne Paris Nord (USPN), dont l'organisme déposant est le Laboratoire Educations et Promotion de la Santé (LEPS) UR3412, représenté par le Pr. Rémi GAGNAYRE, directeur du laboratoire

Investigateur principal : Mme Aude-Marie FOUCAUT, Maitre de Conférence en Sciences et Techniques de Activités Physiques et Sportives, LEPS UR3412, USPN

Investigateur coordonnateur: Mme Albane AUMAITRE, doctorante contractuelle de l'Ecole Doctorale ERASME, LEPS UR3412, USPN

Vous êtes invité·e à participer à une étude interventionnelle se déroulant dans 15 départements de France métropolitaine, en partenariat avec la Ligue Nationale contre le cancer. Celle-ci fait partie d'une thèse doctorale de l'Université Sorbonne Paris Nord, s'adressant à 150 personnes qui ont vécu un cancer, qui ont terminé les traitements contre ce dernier, et qui éprouvent des difficultés – quelles qu'elles soient – à avoir une activité physique régulière. Nous parlons bien ici d'activité physique, et non de « sport ». L'activité physique correspond à toutes les activités où votre corps est en mouvement dans la vie quotidienne, les déplacements, le travail et les loisirs

Objectifs: Cette étude est organisée pour comprendre quels seraient les effets d'une intervention personnalisée mêlant différentes approches, sur votre façon de vous mouvoir ou non au quotidien. Il n'y a ici pas de visée moralisatrice ou compétitive, nous cherchons à vous accompagner selon vos besoins et vos souhaits. L'étude DE FACTO 2 nous permettra *in fine* de concevoir des programmes, prenant au maximum en compte les caractéristiques singulières et les besoins des personnes dans l'après cancer, pour les accompagner vers une vie plus active.

Veuillez lire attentivement ces quelques pages d'information et poser toutes les questions que vous souhaitez aux responsables de l'étude.

Ce document comprend 2 parties : l'information essentielle à votre prise de décision, et le formulaire de consentement.

## Si vous acceptez de participer à cette étude, vous devez savoir que :

➤ L'étude implique de participer à un programme de 12 semaines consécutives, mélangeant :

- une unique séance de pratique d'activité physique en individuel avec un professionnel de l'activité physique adaptée en début de programme ;
- des entretiens motivationnels en individuel menés à distance par téléphone, à raison d'un entretien hebdomadaire en moyenne, selon vos disponibilités et vos besoins, conduits par la doctorante de l'étude Mme Albane AUMAITRE;
- deux ateliers collectifs (10 personnes) de discussion par rapport aux thèmes de l'activité physique et de la sédentarité<sup>1</sup>. Le premier aura lieu en début de programme et le second en fin de programme (avec le professionnel de l'activité physique adaptée

.

<sup>&</sup>lt;sup>1</sup> Temps passé en position assise ou allongée







qui sera intervenu lors de la séance de pratique individuelle). Selon la situation sanitaire, ces ateliers pourront avoir lieu en présentiel ou en distanciel.

- ➤ Vous recevrez une montre connectée qui vous sera laissée à la suite de l'étude. Cette montre recueillera les temps pendant lesquels vous êtes en mouvement ou au repos ;
- ➤ Ce sera à vous de nous mettre à disposition les données vous concernant à l'aide de la montre connectée, procédure dans laquelle nous vous accompagnerons ;
- ➤ Les données recueillies via la montre connectée sont : le nombre de pas, la distance parcourue, l'intensité d'activité physique, le nombre de marches montées, le rythme cardiaque, les cycles de respiration. La montre ne permettra pas de vous géolocaliser et ne sera pas assimilée à votre nom et prénom mais à un code, cela permettra de garantir votre anonymat ;
- ➤ Vous serez amené·e à remplir un questionnaire dans le mois précédant l'intervention à l'occasion d'un entretien, sur ce qui facilite et ce qui freine votre activité physique quotidienne, c'est également là que nous vous fournirons la montre connectée (nous vous aiderons dans cette démarche lors de l'entretien d'entrée dans l'étude). Puis à la suite des 12 semaines d'intervention, nous reviendrons vers vous à 3 reprises pour des courts temps de recueil de données (par exemple, voir si le temps que vous passez à effectuer une activité physique a évolué ou non). Les évaluations seront donc effectuées au début de l'intervention, et à 3 mois, à 6 mois, puis à 1 an après l'intervention.
- ➤ La période totale de votre participation à l'étude est donc de 16 mois (comprenant l'intervention et les temps de mesure). Vous devrez porter la montre le plus souvent possible entre le début de l'intervention, et la dernière mesure, par conséquent pendant ces 16 mois. Les données seront conservées 60 mois après la fin de votre participation pour de potentielles analyses supplémentaires.
- Les données recueillies sont confidentielles et votre anonymat est garanti tout au long du protocole d'étude, et ce même lors de la publication des résultats de la recherche ;
- ➤ A la suite de votre consentement, vous recevrez les dates précises des différentes étapes de l'intervention et des temps de mesures ;
- ➤ Votre participation est volontaire et doit rester libre de toute contrainte. Elle nécessite la signature d'un document exprimant votre consentement ;
- ➤ Vous pouvez toujours contacter l'équipe de recherche si vous avez besoin d'informations complémentaires ;
- ➤ Vous pourrez avoir accès aux résultats de l'étude en contactant Albane AUMAITRE (+33 (0)6 16 88 31 60 ou albane.au@gmail.com) ou Aude-Marie FOUCAUT (+33 (0)1 48 38 76 42 ou audemarie.foucaut@sorbonne-paris-nord.fr).
- ➤ Cette étude est mise en œuvre après évaluation par un Comité de Protection des Personnes qui a fondé son avis sur la cohérence de l'étude, son aspect éthique et le respect de votre anonymat. Le Comité de Protection des Personnes Nord-Ouest 3 a émis un avis favorable le JJ/MM/AAAA. Une copie de l'avis du CPP Nord-Ouest 3 et du résumé de l'étude sera transmise à l'ANSM pour information ;
- ➤ Le promoteur de cette étude a souscrit une assurance de responsabilité civile auprès de la MAIF (n°de police d'assurance : 3649449M) ;







### Pour participer à l'étude vous devez :

- Être majeur∙e ;
- Avoir été diagnostiqué·e d'un cancer du sein, du poumon, du colon-rectum, ou de la prostate ;
- Avoir terminé les traitements de chimio-radio-immunothérapie depuis minimum 1 mois et au maximum 20 ans ;
- Ne pas atteindre les recommandations nationales d'activité physique<sup>2</sup>;
- Passer plus de 7h par jour en position assise ou allongée hors temps de sommeil;
- Pouvoir lire, comprendre et compléter des questionnaires en langue française ;
- Disposer d'un smartphone afin de télécharger une application (Garmin) permettant de synchroniser les données de la montre ;
- Pouvoir utiliser un objet connecté et effectuer des manipulations simples sur ce dernier (enclencher un bouton, charger l'appareil);
- Pouvoir pratiquer une activité physique ;
- Résider en France métropolitaine ;
- Être volontaire pour participer à l'étude ;
- Avoir signé le consentement éclairé ci-joint.

#### Vous ne pouvez pas participer à cette étude si :

- Vous avez été diagnostiqué·e d'un cancer métastatique ;
- Vous avez terminé les traitements de chimio-radio-immunothérapie depuis moins d'un mois à la date du recrutement, ou depuis plus de 20 ans;
- Vous vivez dans un autre pays que la France (y compris ponctuellement);
- Vous êtes dans une situation où aucune activité physique n'est pas possible suite à des contreindications absolues de votre médecin ;
- Vous êtes enceinte ou allaitante ;
- Vous avez moins de 18 ans ;
- Vous êtes majeur·e sous tutelle ou curatelle;
- Vous êtes privé·e de liberté ;
- Posséder une aide pour la locomotion (i.e. béquille);
- Utiliser des traitements influant la pression artérielle, cardiotoxiques (i.e. anthracycline), antidouleurs (substances morphiniques);
- Avoir été diagnostiqué∙e de quelconque anomalie cardiaque.

## Traitement des données :

Les données issues des questionnaires et des montres seront anonymisées (codées : tout ce qui pourrait être sujet à vous identifier sera remplacé par un code comprenant des chiffres et des lettres), puis analysées à l'aide d'un logiciel statistique. A aucun moment de l'étude les montres connectées auront une autre utilisation que la mesure de votre niveau d'activité physique. La géolocalisation sera désactivée, aucun élément ne pourra permettre de vous identifier personnellement. De plus, chaque personne présente au sein de l'équipe de recherche est tenue au secret professionnel. La seule possibilité de divulgation d'une quelconque information serait dans le cas où l'étude serait soumise à une inspection par la commission d'éthique compétente, où l'équipe de recherche serait alors dans

<sup>&</sup>lt;sup>2</sup> Cela revient à <u>ne pas pratiquer</u> d'activité physique à la limite de l'essoufflement au-delà de 30 minutes par jour, 5 jours par semaine. Les recommandations de l'Organisation Mondiale de la Santé (OMS, 2020) sont les suivantes : consacrer au moins 150 à 300 minutes par semaine à une activité d'intensité modérée (ex. marche, jardinage etcetera soit entre 20 et 40 minutes par jour environ) ou pratiquer au moins 75 à 150 minutes d'activité d'intensité élevée (soit entre 10 et 20 minutes par jour environ) ou une combinaison des deux.







l'obligation de transmettre certaines données personnelles mais cela est exceptionnel, et se déroule dans des critères strictes d'anonymat/de sécurité des données [conformément au Règlement Général sur la Protection des Données (RGPD) du 25/05/18]. Le délégué de la protection des données de l'Université Sorbonne Paris Nord, en lien avec cette étude, est Mr BONNET Timothée (dpo@univ-paris13.fr)

Le traitement des données est effectué avec la méthodologie de référence MR001 (recherche dans le domaine de la santé avec recueil du consentement), établie par la Commission Nationale Informatique et Liberté (CNIL), dont l'autorisation est datée au 17/02/2022.

#### Description des risques et bénéfices :

Si vous n'avez pas de contre-indication à la pratique d'activité physique, le risque en termes de santé, est minime et correspond aux risques entraînés par l'activité physique que vous effectuez habituellement. La contrainte de cette étude est de vous rendre disponible aux séances (en présentiel ou en distanciel) et de bien vouloir être sollicité·e et disponible jusqu'à 1 an après l'intervention pour les évaluations.

Vous pouvez vous attendre à retirer des bénéfices personnels du fait de votre participation à l'étude, qui correspondent à ceux entraînés par l'activité physique (plus d'énergie, moins de ruminations, plus de confiance en vous, une meilleure respiration, ...). Sachez aussi que votre participation nous permettra de mieux comprendre comment un programme tel que celui auquel nous vous invitons à participer, peut prendre place sur l'ensemble du pays, grâce aux comités départementaux de la Ligue Nationale contre le Cancer.

## Retrait de consentement :

Votre participation est volontaire et vous avez le droit de retirer votre consentement à participer à l'étude à tout moment, pour quelque raison que ce soit, et sans devoir vous justifier. Si vous retirez votre consentement à l'étude, vous êtes en droit de demander le retrait de vos données. Nous vous demanderons simplement d'en informer Mme Aude-Marie Foucaut et Mme Albane Aumaitre pour une question de gestion des participants.

Si vous participez à cette recherche, nous vous demandons :

- > De collaborer pleinement au bon déroulement de la recherche ;
- ➤ De ne rien masquer comme information au sujet de votre état de santé, de votre activité physique ou de symptômes que vous ressentez.

Contact: Si vous avez besoin d'informations complémentaires, mais aussi en cas de problème ou d'inquiétude, vous pouvez contacter l'équipe de recherche (Albane Aumaitre et Aude Marie Foucaut) par téléphone : +33 (0)6 16 88 31 60 / +33 (0)1 48 38 76 42 ou par mail : <a href="mailto:albane.au@gmail.com">albane.au@gmail.com</a> / <a href="mailto:audemarie.foucaut@sorbonne-paris-nord.fr">audemarie.foucaut@sorbonne-paris-nord.fr</a>







.....

## Formulaire de consentement de participation à l'étude interventionnelle DE FACTO 2

Je soussigné(é), [NOM, Prénom, Comité départemental]

Accepte de participer à la recherche interventionnelle dans les conditions précisées ci-dessus. J'autorise le Laboratoire Educations et Pratiques de Santé UR 3412 (LEPS) de l'Université Sorbonne Paris Nord, 74 rue Marcel Cachin 93017 Bobigny, à procéder un recueil de données me concernant (comme mon activité physique) dans la période allant de 1 mois avant l'intervention, à 1 an après l'intervention dans le cadre de l'étude interventionnelle sur les Déterminants Et Facteurs de l'ACtivité physique après les Traitements en Oncologie (DE FACTO 2).

J'autorise également le LEPS à exploiter mes données anonymisées à des fins non commerciales de recherche scientifique et de communication (interne et externe).

Je suis informé·e que je peux me retirer de l'étude en avertissant Mme Aude-Marie Foucaut (investigateur principal) et Mme Albane Aumaitre (investigateur coordonnateur) sans avoir à me justifier de la raison qui me pousse à prendre cette décision.

Je déclare que j'ai été informé·e sur la nature de l'étude, son but, sa durée, et ce que l'on attend de moi. J'ai pris connaissance du document d'information. J'ai eu suffisamment de temps pour y réfléchir et en parler avec une personne de mon choix si le besoin s'est présenté (entourage, professionnel de santé). J'ai eu l'occasion de poser toutes les questions qui me sont venues à l'esprit et j'ai obtenu une réponse à mes questions. J'ai compris que des données me concernant seront récoltées suite à ma participation à cette étude et que les chercheurs ainsi que le superviseur se portent garant de la confidentialité de ces données.

Je me reconnais être entièrement rempli de mes droits et ne pourrai prétendre à aucune rémunération pour l'exploitation des droits visés à la présente.

J'ai reçu une copie de la lettre d'information et du consentement éclairé.

Albane AUMAITRE Investigateur coordonnateur

NOM, Prénom Paticipant(e) à l'étude DE FACTO 2

Signature, date

Signature, date